CLINICAL TRIAL: NCT03375073
Title: Positive Communication Within Healthcare Team and Clinical Performance: a Prospective, Randomised and Controlled Simulation Trial.
Brief Title: Positive Communication and Clinical Performance in Anaesthetic Care.
Acronym: ComPerf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Pierre ALBALADEJO, Clinical Professor, Anesthesiology and Intensive Care, University Grenoble Alps
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CESAR001
Record Dates: First submitted 2017-11-22; First posted 2017-12-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Positive Communication; Clinical Performance; Anaesthesiology; High Fidelity Simulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, with a 1:1 allocation ratio
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive communication (Experimental): Positive communication during medical transmission
  Interventions: Other: Positive communication during medical transmission
- Non-optimized communication (No Intervention): Medical transmission with non-optimized communication.

INTERVENTIONS:
Other: Positive communication during medical transmission — Use of positive communication for medical transmission to the anaesthetic team who takes over the patient.
  Arms: Positive communication

SUMMARY:
The emotional and cognitive impact of positive communication between caregivers remains uninvestigated. The investigators hypothesize that positive communication during medical transmission can increase clinical performance for managing a subsequent stressful unexpected adverse event.

DETAILED DESCRIPTION:
When caregivers deal with acute stressful adverse events, cognitive overload and negative emotions can impair cognitive abilities and decrease clinical performance. The beneficial effect of positive communication on patients' emotions has widely been studied. However, the emotional and cognitive impact of positive communication between caregivers remains uninvestigated. The primary purpose of this trial is to study the impact of positive communication between anaesthetic teams during medical transmissions on clinical performance for managing a subsequent stressful unexpected adverse event. Secondary outcomes are to study the impact of positive communication on physiological (heart rate variability) and psychological (psychometric scales) levels of stress.

ELIGIBILITY:
Inclusion criteria

Anaesthetic teams composed with :

* 1 resident in anaesthesiology and critical care AND
* 1 anaesthetic nursing student in second year OR 1 anaesthetic nurse graduated less than 5 years ago

Non-inclusion criteria

* Refusal to be videotaped
* No consent to participate
* Anaesthetic nurses working in a paediatric operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Clinical performance of the anaesthetic team | Each anaesthetic team will be involved once in the scenario. The scenario will last about 6 min (transmission not included). Both assessment of clinical performance will be made within 20 weeks of each simulation session
  Clinical performance in a simulated scenario of laryngospasm occurring in a 7 year old child under general anaesthesia. Clinical performance will be scored from 0 to 100 by two independent blinded assessors, using video records and a pre-established scenario-specific checklist. The primary endpoint will be the mean of the two assessments for each performance.

SECONDARY OUTCOMES:
Heart rate variability | Before the scenario (during 5 min), during medical transmission (2 min), during the scenario before the laryngospasm (2 min), during the laryngospasm (4 min), during the debriefing (20 min), after the debriefing (5 min)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Self-reported stress | Before the scenario (at 5 min), after medical transmission (at 7 min), after the scenario (at 13 min), after debriefing (at 33 min)
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).

CONTACTS AND LOCATIONS:
Locations (1):
- University Grenoble Alps, La Tronche, France

REFERENCES:
- [Derived] Bertrand B, Evain JN, Piot J, Wolf R, Bertrand PM, Louys V, Terrisse H, Bosson JL, Albaladejo P, Picard J. Positive communication behaviour during handover and team-based clinical performance in critical situations: a simulation randomised controlled trial. Br J Anaesth. 2021 Apr;126(4):854-861. doi: 10.1016/j.bja.2020.12.011. Epub 2021 Jan 7. PMID 33422288